CLINICAL TRIAL: NCT02828137
Title: Relationships Between Neutrophil-to-Lymphocyte Ratio and Index of Microcirculatory Resistance in ST-segment Elevation Myocardial Infarction Patients Undergone Primary Percutaneous Coronary Intervention
Brief Title: Relation Between NLR and IMR in STEMI Patients
Status: Completed | Type: Observational
Sponsor: Inha University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: INHAUH 2016-06-012
Record Dates: First submitted 2016-06-30; First posted 2016-07-11 (Estimated); Results first posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-06

CONDITIONS: Myocardial Infarction; Death
MeSH Terms: conditions — Myocardial Infarction; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Low NLR group: Neutrophil-to-Lymphocyte (NLR) Ratio < 1.78
- Intermediate NLR group: 1.78 < Neutrophil-to-Lymphocyte (NLR) Ratio < 3.90
- High NLR group: Neutrophil-to-Lymphocyte (NLR) Ratio > 3.90

SUMMARY:
The neutrophil-to-lymphocyte ratio (NLR) has been proven to be reliable inflammatory marker for atherosclerotic process and predictor for clinical outcomes in patients with various cardiovascular diseases. Recent study reported elevated NLR was associated with impaired myocardial perfusion in ST-segment elevation myocardial infarction (STEMI) patients. The investigators sought to determine whether NLR is associated with coronary microcirculation assessed by index of microcirculatory resistance (IMR) in STEMI patients who undergone primary percutaneous coronary intervention (PCI). A total of 123 patients with STEMI underwent successful primary PCI were consecutively enrolled. NLR at admission was calculated, and the patients were divided into three groups according to NLR tertiles. IMR was measured by intracoronary thermodilution-derived method immediately after index PCI.

DETAILED DESCRIPTION:
A total of 123 consecutive STEMI patients who underwent successful primary PCI and coronary physiologic study immediately after PCI were retrospectively enrolled in the study. All patients underwent index PCI between May 2009 and October 2014 at INHA university hospital. The definition of STEMI was determined by the current guidelines.

Complete blood counts, including total and differential WBC counts, were obtained at the time of admission. Total counts of WBC, neutrophils, and lymphocytes were assessed using an automated blood cell counter (XE-2100, Sysmex Inc., Japan). NLR was calculated as the ratio of the neutrophil counts to the lymphocyte counts. All patients were divided into 3 groups according to the NLR tertiles.

The IMR was assessed shortly after primary PCI by using thermodilution-derived method. After successful interventional reperfusion, intracoronary nitroglycerin (100~200μg) was administered and coronary pressure guidewire (Radi Pressure Wire 5, Radi Medical Systems, Uppsala, Sweden) was calibrated outside the patient. The guidewire was equalized at the distal tip of guiding catheter, and then advanced towards the distal third of infarct related artery (IRA). Three times of saline injection (3~5 ml) were administered to IRA and baseline mean transit time was assessed. Microcirculatory hyperemia was induced by using an adenosine infusion (140 μg/kg.min) administered via peripheral venous line. During maximal hyperemia, hyperemic mean transit time (Tmn) was measured using same method as prior separate saline injections. Mean aortic (Pa) and distal coronary pressures (Pd) was measured during hyperemia. The IMR was calculated the formula as follows: IMR = Pd x hyperemic Tmn. Fractional flow reserve (FFR) was calculated by ratio of Pd to Pa during maximal hyperemic status. Coronary flow reserve (CFR) was derived from dividing the resting Tmn by hyperemic Tmn.

Continuous variables were presented as mean ± standard deviation (SD) and categorical variables as the number of patients (percentages). The one way analysis of variance (ANOVA) was used for comparing continuous variables. Additionally, post-hoc analysis was performed for evaluating to be significant by ANOVA. The Pearson's chi-square test or Fisher's exact test was used for analyzing categorical variables. Linear regression analysis was performed for investigating the association between NLR and variables using clinical, laboratory, echocardiographic, and angiographic data. A p value <0.05 was regarded statistically significant. All statistical analyses were carried out with SPSS version 19.0 (SPSS inc., Chicago, Illinois, USA).

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients who undergone primary PCI

Exclusion Criteria:

* unprotected left main coronary artery disease
* stent thrombosis presentation
* a history of coronary artery bypass graft surgery
* prior intravenous thrombolytic therapy before PCI
* high degree atrioventricular block
* remained cardiogenic shock after complete PCI
* contraindication for use of adenosine
* post-PCI thrombolysis in myocardial infarction (TIMI) flow grade 0 or 1

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 123 consecutive STEMI patients who underwent successful primary PCI and coronary physiologic study immediately after PCI were retrospectively enrolled in the study. All patients underwent index PCI between May 2009 and October 2014 at INHA university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2009-05; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided
If it is feasible to upload the individual data, the investigator would consider it positively.

REFERENCES:
- [Derived] Lee MJ, Park SD, Kwon SW, Woo SI, Lee MD, Shin SH, Kim DH, Kwan J, Park KS. Relation Between Neutrophil-to-Lymphocyte Ratio and Index of Microcirculatory Resistance in Patients With ST-Segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention. Am J Cardiol. 2016 Nov 1;118(9):1323-1328. doi: 10.1016/j.amjcard.2016.07.072. Epub 2016 Aug 13. PMID 27600462

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low NLR Group | Intermediate NLR Group | High NLR Group
Started | 41 | 41 | 41
Completed | 41 | 41 | 41
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low NLR Group | Intermediate NLR Group | High NLR Group | Total
Number analyzed (Participants) | 41 | 41 | 41 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 32 | 30 | 96
  >=65 years | 7 | 9 | 11 | 27
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 55 (10) | 55 (11) | 58 (12) | 57 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 3 | 13
  Male | 35 | 37 | 38 | 110
Region of Enrollment [Number; unit: participants] — Incheon Province in the Western part of South Korea
  participants
    Korea, Republic of | 41 | 41 | 41 | 123

OUTCOME MEASURES:

1. Primary Outcome: Index of Microcirculatory Resistance
Description: IMR in low NLR group : 21.94 ± 12.87 IMR in intermediate NLR group : 23.22 ± 12.73 IMR in high NLR group : 32.95 ± 20.60
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: IMR
Groups:
- Low NLR Group: Neutrophil-to-Lymphocyte (NLR) Ratio < 1.78 IMR 21.94 ± 12.87
- Intermediate NLR Group: 1.78 < Neutrophil-to-Lymphocyte (NLR) Ratio < 3.90 IMR 23.22 ± 12.73
- High NLR Group: Neutrophil-to-Lymphocyte (NLR) Ratio > 3.90 IMR 32.95 ± 20.60
Arm/Group | Low NLR Group | Intermediate NLR Group | High NLR Group
Number analyzed (Participants) | 41 | 41 | 41
IMR | 21.94 (12.87) | 23.22 (12.73) | 32.95 (20.60)

ADVERSE EVENTS:
Arm/Group | Low NLR Group | Intermediate NLR Group | High NLR Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No